CLINICAL TRIAL: NCT04600427
Title: Epidural Blockade for Ogilvie's Syndrome: A Prospective Pilot Study
Brief Title: Epidural for Ogilvie's Syndrome
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This was a pilot study aimed at assessing feasibility of further assessing epidural as a treatment for Ogilvie's. There were no eligible patients that were enrolled throughout the two years of accrual. Thus we deemed the study not feasible.
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12731
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2021-09

CONDITIONS: Ogilvie Syndrome; Colonic Pseudo-Obstruction
MeSH Terms: conditions — Colonic Pseudo-Obstruction | interventions — Anesthesia, Epidural

STUDY DESIGN:
Intervention Model Description: Single arm, single centre study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Epidural anesthesia (Experimental): The patient will be positioned appropriately and the T11-12 (if not accessible we will accept 1-2 spaces above or below) interspace landmarked using established ultrasound guidance techniques. The patient's back will be prepped and draped in a sterile fashion. An epidural catheter will be inserted into the T11-12 interspace with a midline or paramedian approach using a 17G Tuohy needle. Plain preservative free bupivicaine 0.25% will be the local anesthetic used. After a 2-3 mL test dose to rule out intrathecal catheter positioning, a loading dose of 5-8 mL will be administered over 5-10 minutes to further rule out intravascular positioning of the catheter. Successful epidural placement will be defined by catheter insertion and confirmed by sensory blockade assessed by ice or pin prick testing. When correct positioning is confirmed, a continuous infusion of 3 mL per hour of bupivacaine 0.25% plain solution will begin.
  Interventions: Procedure: Epidural anesthesia

INTERVENTIONS:
Procedure: Epidural anesthesia — T11-12 epidural blockade with 0.25% bupivacaine continuous infusion.

SUMMARY:
Epidural anesthesia may represent a safe and effective pharmacological tool in the management of Ogilvie's Syndrome. This pilot study aims to demonstrate feasibility, safety, and efficacy of epidural anesthesia to set the stage for adequately powered future randomized controlled trials (RCTs) in order to assess the efficacy of epidural anesthetic as a pharmacological treatment strategy for Ogilvie's Syndrome. Ultimately, this research may prompt further investigation and establish standardized criteria for managing Ogilvie's Syndrome patients with epidural anesthesia.

DETAILED DESCRIPTION:
Currently, treatment pathways for Ogilvie's Syndrome suggest observation and attempted correction of the potential precipitating factors for 24 to 72 hours following radiologic assessment if the cecum is less than 12cm and abdominal imaging does not demonstrate signs of impending perforation. Should symptoms fail to resolve beyond 72 hours, and the cecum remain under 12cm without worsening clinical status, pharmacologic intervention with neostigmine is indicated. Symptoms resolve in 60% to 90% of patients following administration of single dose of neostigmine, however continued monitoring is required as up to 40% of these patients can experience recurrent colonic dilation. Additionally, neostigmine can be associated with serious adverse events such as bradycardia and bronchospasm. Altogether, there may be potential for further optimization of the pharmacologic management of Ogilvie's Syndrome.

Given the predominant theory that Ogilvie's Syndrome is caused by sympathetic overdrive, the splanchnic sympathetic blockade provided by epidural anesthesia could be of theoretical benefit. In 1988, a small, prospective cohort study evaluated the use of epidural anesthesia in eight patients with Ogilvie's Syndrome. Symptoms were controlled and cecal dilation resolved without recurrence in 62.5% of these patients, and the authors concluded that with further study, the use of epidural anesthesia could be a reasonable alternative to neostigmine. Yet, no subsequent studies were performed.

This proposed single-arm, single-center prospective cohort pilot study will examine the feasibility, safety, and efficacy of epidural anesthesia in patients with Ogilvie's Syndrome refractory to conservative management. Adult patients with a documented diagnosis of Ogilvie's Syndrome admitted as an inpatient to St. Joseph's Healthcare Hamilton (SJHH) who failed conservative management will be included. Following assessment of eligibility and the informed consent process, patients will be evaluated by the acute pain service anesthesiologist. A low-dose bupivacaine (0.25%) infusion will commence following insertion of an epidural catheter at the T11-12 interspace, with a loading dose of 5-10mL followed by a 3mL per hour infusion. Monitoring for resolution of disease will take place iteratively by the general surgery team, and failed symptom resolution will mandate further treatment in the form of colonoscopic decompression or surgical intervention. Patients will be followed throughout their index hospital and stay and up to 30 days following discharge from hospital. Feasibility will be assessed through recruitment rate and rate of successful epidural placement. The rate of epidural anesthesia-related morbidity within 30 days of treatment will serve as the primary safety measure. The primary efficacy measure is clinical and radiologic resolution without recurrence.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Admitted to an inpatient ward at SJHH with a documented diagnosis of Ogilvie's Syndrome/Acute Colonic Pseudo-Obstruction
* Failed conservative management for at least 24-48 hours

Exclusion Criteria:

* Hemodynamic instability
* Peritonitis on abdominal examination
* Cecal diameter greater than 12cm or evidence of hollow viscus perforation on abdominal imaging (e.g. bowel wall thickening, mesenteric stranding, hypoenhancement of bowel wall)
* Documented allergic reaction to anesthetic agent
* Bacteremia
* Local soft tissue infection at the puncture site
* Coagulopathy or therapeutic anticoagulation
* Intracranial pathology leading to increased intracranial pressure
* Prior spinal surgery
* Unstable severe respiratory or cardiovascular disease
* Previously managed with epidural anesthesia for Ogilvie's Syndrome
* Inability/unwilling to consent to trial treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 2 years
  Larger study will be considered feasible if a recruitment rate of 1 patient per month is achieved.
Successful epidural insertion | 2 years
  A minimum successful epidural insertion rate of 80%. Successful epidural placement will be defined by catheter insertion and confirmed by sensory blockade assessed by ice or pin prick testing.
Follow-up rate | 2 years
  Larger study will be considered feasible if more than 80% of patients recruited have a full 30 days of follow up data.
Epidural-related morbidity | 30 days
  . Overall morbidity will include the following complications: hypotension, nausea, vomiting, bronchoconstriction, post dural-puncture headache, transient neurological syndrome, neurologic deficit, meningitis, epidural hematoma, epidural abscess, osteomyelitis, and systemic local anesthesia toxicity.
Rate of clinical resolution | 2 years
  Clinical resolution will be defined as passage of flatus and stool with associated resolution of abdominal distention and bloating.
Rate of radiological resolution | 2 years
  Radiological resolution will be defined as decreased cecal diameter to less than 9cm

SECONDARY OUTCOMES:
Readmission rate | 30 days
  Rate of readmission to hospital following intervention and subsequent discharge will be reported as secondary safety outcomes.
Length of stay in hospital | 30 days
  Length of stay in hospital following placement of epidural anesthesia
Mean time to clinical resolution | 2 years
  Clinical resolution will be defined as passage of flatus and stool with associated resolution of abdominal distention and bloating.
Mean time to radiological resolution | 2 years
  Radiological resolution will be defined as decreased cecal diameter to less than 9cm

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Healthcare, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No